CLINICAL TRIAL: NCT06875089
Title: A Pilot Study to Assess the Feasibility and Acceptability of Newborn Screening Using in Silico Panel-based Solo Genome Sequencing in France PERIGENOMED-CLINICS 1 (PGC1 Study)
Brief Title: A Pilot Study to Assess the Feasibility and Acceptability of Newborn Screening Using in Silico Panel-based Solo Genome Sequencing in France
Acronym: PGC1
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: OLIVIER FAIVRE AFM 2023
Record Dates: First submitted 2025-02-26; First posted 2025-03-13 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Newborn Screening Programmes for Rare Diseases
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No participants: future families not taking part in the pGS- NBS study
  Interventions: Other: Satisfaction questionnaire; Other: interview with HSS researcher
- Participants: future families who take part the pGS-NBS
  Interventions: Genetic: pGS-NBS; Other: Satisfaction questionnaire; Other: interview with HSS researcher; Other: Qualitative and quantitative longitudinal exploration; Other: Medical follow up

INTERVENTIONS:
Genetic: pGS-NBS — Collection of a second DBS card if the parents accept the pGS-NBS for their newborn
  Groups: Participants
Other: Satisfaction questionnaire — questionnaire on information process of parents informed about pGS-NBS
Other: interview with HSS researcher — interview with a member of the HSS team on reasons for declining /accepting pGS-NBS
Other: satisfaction questionnaire — questionnaire on results delivery in parents having accepted the pGS-NBS
  Groups: Participants
Other: Qualitative and quantitative longitudinal exploration — validated anxiety and depression scales to assess the psychosocial impact and perceived utility for families whose child screened negative among which 30 families will be interviewed. Interviews and validated anxiety and depression scales will be suggested to all families receiving positive screening results
  Groups: Participants
Other: Medical follow up — follow-up of true positives and false negatives based on medical records (vital status, care pathways) until 5 years after results delivery
  Groups: Participants

SUMMARY:
Newborn Screening (NBS) based on genome sequencing (GS) is currently the subject of particular attention at both European and international levels. Over the past three years, several publications have discussed the opportunities and challenges of using GS for NBS. To date, only two Chinese programs have published their results, the first on a series of 29,601 healthy newborns and the second on a series of 10,334 healthy newborns and 668 high-risk infants. Globally, more than twenty pilot projects are underway, although none has been initiated within the French context thus far. Across the different pilot projects, various study designs are used. Most have opted for a targeted GS-based analysis to screen for pediatric-onset diseases. Some projects focus solely on diseases for which effective drugs or interventions exist to prevent or reduce symptoms. In contrast, others offer parents the option to screen their newborns for diseases without current treatment options, but for which a treatment is underdevelopment, or with interest in early management, a choice exercised by most parents. Indeed, early diagnosis of these diseases can help to introduce treatments or interventions when they become available, to participate in research trials on new treatments and to receive early management and genetic counseling.

In France, the national NBS program has long been recognized worldwide for its organizational quality and comprehensiveness, although, until recently, it has one of the lowest numbers of diseases screened in Europe. As of mid-2024, the French NBS only includes 14 serious diseases. Recently, the French bioethics law has evolved to allow the use of genetic testing as a first-line procedure for NBS. At the same time, the development and efficiency of genomic techniques and the rapid increase in the number of treatable rare diseases (RDs) raise questions about the acceptability and relevance of these genomic methods for NBS and its possible extension. The extension of NBS to many RDs of early onset represents a real public health challenge as RDs, 80% of which are of genetic origin, account for 10% of deaths before the age of 5.

The FHU TRANSLAD has elaborated the PERIGENOMED Project, a large-scale project which aims to assess the relevance of pGS-NBS in France (analytical and clinical validity, clinical utility and psychosocial, ethical and organizational issues).

The pGS-NBS (also known as in silico panel-based GS, i.e. an analysis carried out entirely using informatic tools) consists of bioinformatics filtering steps that return only selected variants and/or rare variants from targeted genes issued from GS. So, even if the source data comes from the GS, it is possible to configure the pipeline to return only those variations known to be responsible for specific RDs.

the PERIGENOMED Project will be led in two steps. The first pilot step (PERIGENOMED-CLINICS 1 - PGC1 Study), presented in this protocol, aims to evaluate the feasibility and acceptability of pGS-NBS France. This pilot study plans to screen 2,500 newborns using pGS-NBS targeting two lists of genes (1 corresponding to genes variables responsible of treatable rare diseases, 2 including genes variation leading to actionable rare diseases). In both lists only RDs of early onset are considered. PGC1 study will be carried in 5 healthcare centers in France, with results expected to be returned to clinicians within less than 4 weeks. It will also provide an understanding of the optimal information and analytical pathways, and the possible organizational repercussions of pGS-NBS as well as a first insight about the validity of the pGS-NBS and about the clinical course of newborns screened positive and with a confirmed RD Two studies in humanities and social sciences (HSS) will also be linked to PGC1 Study. The first will focus on the reasons given by decliners and on the medical and socio-economic characteristics (at the individual and contextual level) of decliners versus participants. The second will assess the psychosocial impact of result disclosure on families of positive newborns, comparatively of negative ones.

These initial results will provide the first outcomes before the launch of a second larger phase PERIGENOMED-CLINICS 2 (PGC2 Study - 22,000 newborns), designed for studying the implementation of such pGS-NBS in routine on a regional level.

ELIGIBILITY:
Inclusion Criteria:

For satisfaction study about the information & identification of determinants of acceptability :

Inclusion criteria for parents/legal guardians :

* All future parents approached for whom the unborn child will be cared for in the participating maternity unit
* At least one parent/legal guardian who received information about the study
* Future parents/legal guardian who do not object to the use of their data
* Parent(s) or legal guardian(s) affiliated to a social security system or beneficiaries of such a system

For pGS-NBS :

Inclusion criteria for newborn :

* All babies born in one of the participating centers or born by chance outside the maternity but whom care will be carried out in the participating center
* Newborn who are less than 28 days at the date of the collection of PGC1 blotting paper

Inclusion criteria for parents/legal guardians

* At least one biological parent who received information about the study
* Parent(s) or legal guardian(s) who do not object to "conventional" NBS
* At least one parent/legal guardian able to provide consent for testing the infant
* Informed consent signed by at least one parent/legal guardian
* Agreement of the second parent/legal guardian for testing the infant (unless he is unknown or loss of contact) obtained from the first parent/legal guardian if his written informed consent has not been obtained
* Parent(s) or legal guardian(s) affiliated to a social security system or beneficiaries of such a system

Exclusion Criteria:

Non inclusion criteria for satisfaction studies and pGS-NBS :

Non-inclusion criteria for parents/legal guardians :

* Parent(s) or legal guardian(s) under legal protection (guardianship, tutorship) or to a court order Non-inclusion criteria for newborn
* Babies born under anonymous birth according to the French law, known as "nés sous X"

Ages: 0 Days to 28 Days | Sex: All
Age Groups: Child
Study Population: all the parents of live newborns in each participating maternity unit
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
parents who have accepted the pGS-NBS for their children for Treatable list | until 2 days after birth with extension up to 28 days in case of hospitalization in intensive care
  number of families taking part the pGS-NBS (Treatable list) among the families who were offered the pGS-NBS in the centers over the inclusion period. If this number is at least of 603/1251, we will be able to reject that the percentage of acceptance is below 45% versus the alternative that it is greater Conversely, if the number is equal or below 602/1251, we will reject the hypothesis that the acceptability is at least 50%.
results concerning the Treatable list returned to clinicians within 4 weeks following the sample | 4 weeks following the sample
  number of families for which the pGS-NBS results concerning the Treatable list are delivered to clinicians in less than 4 weeks among those who consent to the pGS-NBS. If this number is at least 219/220, we will reject our null hypothesis (i.e. that the feasibility rate is less than or equal to 95% versus the alternative hypothesis that it is greater).

SECONDARY OUTCOMES:
parents who have accepted the pGS-NBS for their children for Actionable list | until 2 days after birth
  percentage of families taking part to the pGS-NBS based on the complementary list of genes (Actionable list) among the families who were offered the GS NBS in the centers over the inclusion period
results concerning the Actionable list returned to clinicians within 4 weeks following the sample, | 4 weeks following the sample
  Results concerning the Actionable list returned to clinicians, 4 weeks following the sample organizational indicators constributing to the feasibility assessment of the pGS-NBS : duration of analytical processes, human resources, technical difficulties, screenings requiring a 2nd sample,
Questionnaire for parents' satisfaction with the screening and reporting processes | up to 4 weeks
  (flash questionnaire for all parents and complementary questionnaire for parents who accept it)
profiles of parents who take part or not to pGS-NBS | at the baseline
  Interviews
quantitative exploration | At : 1,6,12,24,36,48 and 60 months after positive results delivery At : 1 and 12 months after negative results delivery
  anxiety and depression scales
pGS-NBS performance | 5 years;
  Children with negative results identified as false negative by reference centers and/or NDBRD (National Data Bank for Rare Diseases) before age 5
Clinical evoluation of newborns with true positive results until 5 years | 5 years
  medical observations up to age 5 (collection of follow-up as part of standard care) of newborns with positive results
pGS-NBS performance | 3 months post pGS-NBS results delivery
  Children with positive results with pGS-NBS not confirmed by the diagnostic assessment
pGS-NBS performance | frame 1 month after the birth
  Identification of one of the 14 diseases in the conventional NBS
qualitative exploration | At : 1,6,12,24,36,48 and 60 months after positive results delivery At : 1 and 12 months after negative results delivery
  interviews

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - CHU d'Angers, Angers
  - CHU Besançon, Besançon
  - CHU Dijon Bourgogne, Dijon
  - CHU Hôtel Dieu, Nantes
  - CHU Rennes - Hôpital Sud, Rennes

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Level C, Thauvin-Robinet C, Binquet C, Duffourd Y, Davoine E, Chevarin M, Tran-Mau-Them F, Lemaitre M, Bruel AL, Safraou H, Salvi D, Tisserant E, Lecommandeur E, Charreton A, Hassine A, de Tayrac M, Redon R, Barc J, Schmitt S, Piard J, Kuentz P, Cormier C, Malbos M, Racine C, Chabrol B, Cheillan D, Tardy V, Colin E, Bris C, Mercier S, Nizon M, Gaudillat L, Loizeau V, Lenelle C, Mottet N, Simon E, Arnoux JB, Carpentier M, Renaud C, Ziegler A, Lejeune C, Jannot AS, Asensio ML, Rollier P, Odent S, Bezieau S, Pasquier L, Huet F, Faivre L. PERIGENOMED-CLINICS 1-the first study on feasibility, acceptability and psychosocial impact of PERIGENOMED: a pilot project aimed at providing initial concrete evidence on the relevance of panel-based genome sequencing for newborn screening (NBS) in France. BMJ Open. 2025 Oct 23;15(10):e105752. doi: 10.1136/bmjopen-2025-105752. PMID 41130699